CLINICAL TRIAL: NCT05101525
Title: Study of the Functional Result of the Reinsertion of the Subscapular in Reverse Shoulder
Brief Title: Study of the Functional Result of the Reinsertion of the Subscapular in Reverse Shoulder Prostheses According to the Healing of the Subscapular
Acronym: CICASCAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A01483-54
Record Dates: First submitted 2021-10-28; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Reverse Shoulder Prothesis; Healing of the Subscapularis
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with effective tendon healing (Experimental)
  Interventions: Procedure: Ultrasound
- Patient without tendon healing (Active Comparator)
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound to visualize the intra tendinous marker. If this is in place, healing is effective. On the other hand, if it has migrated, there is no scarring.

SUMMARY:
This study is based on the hypothesis that the functional result is better if the subscapularis is reinserted and healed. The originality of the study therefore consists in systematically monitoring the healing of this tendon postoperatively, with sufficient follow-up, by ultrasound and by an intra-tendon marker, in order to differentiate the result depending on whether the tendon is healed or not.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 years old
* Patient with an indication of reverse prosthesis for cuff rupture, or eccentric omarthrosis, or omarthrosis without cuff rupture but with posterior eccentricity
* Patient with a normal subscapularis preoperatively
* Patient benefiting from a social protection insurance
* Patient having signed the free and informed consent

Exclusion Criteria:

* Patient with an indication of anatomical prosthesis
* Patient with an abnormal subscapularis preoperatively
* Patient operated for a revision of prosthesis
* Patient with an indication for prosthesis on fracture sequelae
* Patient with an indication for prosthesis on fracture
* Patient participating in another clinical study
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, breastfeeding or parturient woman
* Patient hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-03-09 (Estimated); Study Completion 2025-03-09 (Estimated)

PRIMARY OUTCOMES:
Mobility of internal rotation evaluation | 12 months
  The mobility of internal rotation will be assessed with the level of medial rotation of the Constant score (0 to 100 points - 5 different themes - 11 items)
Tendon healing assessment | 12 months
  The healing will be evaluated by an ultrasound allowing to visualize the intra tendinous marker. If this is in place, healing is effective. On the other hand, if it has migrated, there is no scarring

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Martin Private Hospital, Caen, Normandy, France